CLINICAL TRIAL: NCT04634006
Title: The Acute and Long-Term Effect of Home-Based Transcranial Direct Current Stimulation on Clinical Symptoms and Executive Function in Children With ADHD: A Randomized, Sham-Controlled tDCS and fNIRS Study
Brief Title: Home-Based tDCS in Children With ADHD: A Randomized, Sham-Controlled tDCS and fNIRS Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Choi Deblieck, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/056
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Attention Deficit Disorder (ADD)
Keywords: tDCS; fNIRS; home-based; Executive functioning; Attention; Inhibitory control; DLPFC; IFG; Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, parallel assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- active tDCS 1 (Active Comparator): Anodal tDCS will be applied over the left DLPFC (F3) according to the 10-20 EEG electrode systems and the cathode will be placed over the the vertex (Cz), using square saline-soaked sponge pads 25 cm2. The current intensity of 1 mA will be used for 20 mins for a session. (N=25)
  Interventions: Device: Home-based transcranial direct current (tDCS) device
- active tDCS 2 (Active Comparator): Anodal tDCS will be applied over the right IFG (1/3 of the distance between F8 and C6) according to the 10-20 EEG electrode systems and the cathode will be placed posterior to left mastoid, using square saline-soaked sponge pads 25 cm2. The current intensity of 1 mA will be used for 20 mins for a session. (N=25)
  Interventions: Device: Home-based transcranial direct current (tDCS) device
- sham tDCS (Sham Comparator): Anodal tDCS will be applied over the left DLPFC (N=13) or right IFG (N=12) according to the 10-20 EEG electrode systems and the cathode will be placed over vertex or posterior to left mastoid, respectively, using square saline-soaked sponge pads 25 cm2. Sham stimulation will be maintained for 19 min without current flow by increasing current for 30 s followed by a decrease for 30 s.
  Interventions: Device: Home-based transcranial direct current (tDCS) device

INTERVENTIONS:
Device: Home-based transcranial direct current (tDCS) device — tDCS is a brain electrostimulation technique that consists of applying a current of low intensity (between 1 and 2 mA) on the scalp via two electrodes in order to modify the cerebral activity of the stimulated zones. Twenty sessions (active/sham) will be self-administered by parent or caregiver on twenty consecutive business days. The parameter of electrode size, current strength and current duration were previously tested for safety in children. The investigators use the Soterix Medical tDCS devices of the home-based miniCT 1x1 type.

SUMMARY:
The purpose of this study is to investigate the efficacy of twenty daily sessions of home-based tDCS over the left DLPFC, right IFG on attention and response inhibition in children with ADHD. Investigators hypothesize that multiple sessions of tDCS will induce a greater and long-term effect on attentional and/or inhibitory response in children with ADHD. In addition, this study seeks to get a better understanding of the mechanisms of tDCS using fNIRS.

DETAILED DESCRIPTION:
BACKGROUND: Attention deficit/hyperactivity disorder (ADHD) is one of the most impairing neurodevelopmental disorders of childhood with a worldwide prevalence of 5.3% in children. It is featured by the presence of a persistent pattern of inattention and/or hyperactivity-impulsivity that profoundly affects or reduces the quality of social, academic, and occupational achievements. Influential models of ADHD mainly focus on a deficit in inhibitory control that leads to executive dysfunctions, associated to neural alteration in the prefrontal areas, the striatum, and the cerebellum. Although ADHD can be effectively treated with psychostimulants, a significant proportion of patients discontinue treatment because of adverse events or insufficient improvement of symptoms. In addition, cognitive abilities that are frequently impaired in ADHD are not directly targeted by medication. Therefore, additional treatment options, especially to improve cognitive abilities, are needed. Because of its relatively easy application and well-established safety, non-invasive brain stimulation, such as transcranial direct current stimulation (tDCS), is a promising additional treatment option for children with ADHD. To date, only eight studies have submitted children with ADHD to a maximal of 5 daily sessions. The fact that the technology is inexpensive, and has the potential of being used as a portable device at home by patients, further renders tDCS an attractive tool to explore in treatment in children with neuropsychological disorders, including ADHD. Further, functional near infrared spectroscopy (fNIRS), a non-invasive, compact, unrestrictive, and accessible functional neuroimaging modality has demonstrated its potential in the clinical diagnosis of ADHD children. Since fNIRS visualizes the neural attention and inhibition processes in children with ADHD while they perform tasks online, this technique may have great potential in recording neural changes by tDCS.

OBJECTIVES: The investigators aim to explore the acute and long-term effect of 20 daily sessions of home-based tDCS while doing homework. Our primary objectives seek to determine if tDCS improves: 1) ADHD symptoms, 2) executive function and/or inhibitory processes in children with tDCS. Our secondary aims look at 1) depressive and anxiety symptoms in children with ADHD and 2) the safety and feasibility of home-based tDCS in children with ADHD, and 3) evaluate the mechanisms through which tDCS could be therapeutic using fNIRS that reveals neuroplastic changes successfully.

METHODS: 75 children with ADHD will be submitted to a home-based active or sham fixed-dose tDCS (20 minutes of 1 mA) in a 1:1:1 double-blind, sham-controlled, randomized, parallel-group scheme. Children will be randomly assigned to receiving either 1) active tDCS of anodal left DLPFC and cathodal vertex, 2) active tDCS of anodal right IFG and cathodal posterior to left mastoid or 3) sham tDCS. Stimulation sessions will occur daily, Monday through Friday, for 20 days over a 4-week period. To determine the acute and longterm efficacy of home-based tDCS, children, parents, and teachers will be asked to weekly fill in questionnaires and/or perform tasks online on the weekend from their home. 1) ADHD symptoms will be evaluated using ADHD, DBD and VAS scales. Executive function and inhibitory processes will be determined by a change in I) Visual Search Task, II) Stroop Task, III) Go/No Go Task, IV) Stop Signal Task. 2) Depression/anxiety symptoms will be assessed using HADS and IDS-C scales. Safety and feasibility of home-based tDCS will be assessed using VAS scales and an adverse events questionnaire. Lastly, a change in oxygenated hemoglobin and deoxygenated hemoglobin will help elucidate the mechanisms of tDCS on ADHD. After the tDCS intervention, children will be asked to stay medication-free for as long as they can until study completion for maximal 1-month-post tDCS. All children will be evaluated in person at baseline (visit 1), immediately after the 4-week-treatment (visit 2), and a last visit within 1 month after treatment (visit 3). During these three visits, brain activation patterns of the children will be assessed online using fNIRS while performing the four behavioral tasks.

CONCLUSION: This study will be the first to increase the number of daily sessions of tDCS from 5 to 20 in children with ADHD, making it more than 5 times more likely to increase the response rate to tDCS. Knowledge gained by non-invasive brain stimulation (NIBS) research in children with ADHD might be translatable into an alternative effective treatment, reduce side-effects, and advance the development of closed-loop neuromodulation in ADHD in general. Additionally, no home-based remote tDCS study has ever been conducted in children. Demonstrating its potential will not only offer a more feasible alternative to daily laboratory visits or clinical consultations but may also reduce patient and clinic costs. Lastly, this study will be the first combining fNIRS and tDCS in order to elucidate the acute and longterm mechanisms of effective tDCS intervention in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-12,
2. ADHD without comorbid conduct disorders, autism or tic disorders as diagnosed according to guidelines by an experienced child and adolescent psychiatrist,
3. Medication satisfaction VAS (<6/10),
4. Sufficient compliance of the child and his/her family,
5. Combined or hyperactive-impulsive type according to DSM-V (American Psychiatric Association 1994)] or for the hyperkinetic disorder according to ICD-10 (F90.0, International Classification of Diseases (ICD), 2010),
6. Right-handed

Exclusion Criteria:

1. Intelligence Quotient (IQ) <80,
2. Other neuropsychiatric or pediatric disorders,
3. Epilepsy, including pathological Electroencephalography-patterns (e.g., increased neural excitability), former cerebral seizure, drug abuse, increased intracranial pressure, former craniocerebral injury accompanied by loss of consciousness,
4. Any metallic implantations in the facial or skull area, cochlear implant, pacemaker.
5. History of exposure to tDCS in the past (to minimizing risk of unblinding sham condition).
6. History of exposure to Electroconvulsive therapy in the past.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder (ADHD) - Parents | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  The questionnaire, a standardized instrument to diagnose ADHD, provides a severity score for each ADHD symptom, and is characterized by psychometric properties that allow detection of changes even in the very brief window of time such as only 1 week. Usually, 0 means never, and 3 or 4 means very often and the higher the score, the more severe the symptom.
Disruptive Behavior Disorders Rating (DBD) - Parents | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  The Disruptive Behavior Disorder rating scale is designed to aid in the diagnostic process for a number of child psychopathologies, particularly externalizing disorders, including the three disruptive behavior disorder categories (Conduct Disorder, Oppositional Defiance Disorder and Attention Deficit Hyperactivity Disorder). Each item is rated on a four-point scale ranging from not at all (0) to very much (3).
Visual Analogue Scale (VAS) - Teachers | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Scores are recorded by stopping the slider on a 10-cm line that represents a continuum between "absent" and "present."Teachers will also be asked to weekly complete horizontal VAS on attention, work independence, motor unrest, impulsivity, keeping appointments, order, playground behavior.
Visual Search - Child | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  Visual Search a measures a conjunction visual search process. Reaction time (RT) and accuracy are dependent on the distractor-ratio and the number of distractors present.
Stroop Task - Child | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  The Stroop task is measure of interference control. The proportion of false answer and reaction time of third stage as the main stage that shows interference stimuli was calculated to assess the interference inhibition.
Go/No Go Task - Child | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  The Go/No Go Task is a measure of prepotent response inhibition. The correct response to No-Go stimuli assesses the prepotent response inhibition in a way that they have to refrain from pressing the arrow button when they see a Stop sign with delay.
Stop Signal Task - Child | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  The Stop Signal Task is another measure of inhibition of prepotent responses. The stop signal reaction time (SSRT), a measure of inhibition, is estimated based on the notion of a race between a go process, which is triggered by the presentation of the go stimulus, and a stop process, which is triggered by the presentation of the stop signal.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of home-based tDCS in children with ADHD | From Start to treatment termination
  Frequency of premature study terminations between patients randomized to tDCS versus those randomized to sham treatment, the safety of tDCS by comparing the severity and frequency of serious adverse events (AEs), treatment-emergent AEs, and total AEs during each visit, the number of days the child/parents decide to stay medication free post tDCS treatment for maximal 1 month will also be carefully recorded. Children and parents will also report feasibility using a visual analogue scale (VAS).
Hospital Anxiety and Depression Scale (HADS) - Children | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  To evaluate the effect of home-based tDCS on secondary ADHD symptoms, i.e., depression and anxiety, in children with ADHD. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Inventory of Depressive Symptomatology Clinician (IDS-C) - Parents | Change form baseline to week 1 to week 2 to week 3 to week 4 to 1 week post treatment to 1 month post treatment
  To evaluate the effect of home-based tDCS on secondary ADHD symptoms, i.e., depression and anxiety, in children with ADHD. The IDS-C total scores range from 0 to 27. The total score is obtained by adding the scores for each of the nine symptom domains of the DSM-IV Major Depressive Disorder criteria: depressed mood, loss of interest or pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, and psychomotor changes. Each item is rated 0-3.
Hemodynamic Response | Baseline to 1 Week post tDCS to 1 Month Post tDCS
  Changes in oxygenated hemoglobin (oxy-Hb), deoxygenated hemoglobin (deoxy-Hb), and total hemoglobin (total-Hb) concentration changes will be calculated with the modified Beer-Lambert Law using the NIRSIT-Lite Kids functional Near-Infrared spectroscopy device made by OBELAB Inc. The device radiates a Light Emitting Diode (LED) light with an output of 1 milliwatt (mW) or less which is harmless to the human body. The device comes with PC software that can be used to monitor the distribution of cerebral oxygen saturation via multiple channels (OBELAB Inc.).

CONTACTS AND LOCATIONS:
Overall Officials: Choi Deblieck, PhD, Principal Investigator — UPC KU Leuven; Liesbet Devalkeneer, MD, Principal Investigator — OLVZ Asse
Locations (1):
- OLVZ Asse, Asse, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No